CLINICAL TRIAL: NCT05078333
Title: Comparison of Effectiveness of Dry Needling and High Intensity Laser Therapy in Treatment of Myofascial Pain Syndrome: A Randomized Single-blind Controlled Study
Brief Title: Dry Needling and High Intensity Laser Therapy in Treatment of Myofascial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emine Dundar Ahi (Other)
Responsible Party: Sponsor-Investigator, Emine Dundar Ahi, Principal Investigator, Kocaeli University
Organization: Kocaeli University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K-064
Record Dates: First submitted 2021-09-20; First posted 2021-10-14 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Myofascial Pain Syndrome
Keywords: Myofascial pain syndrome; high-intensity laser therapy; dry needling; exercise
MeSH Terms: conditions — Myofascial Pain Syndromes; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- exercise (No Intervention): All patients in all three groups will perform 15 sessions (for 3 weeks, weekdays), cervical area isometric strengthening exercises, active ROM exercises and stretching exercises for 15 minutes a day with the same physiotherapist.
- exercise+HILT (Active Comparator): In addition to the exercise program, randomly selected 36 case patients + HILT (BTL brand 6000 series, United Kingdom), to the cervical area, for the a period of 3 week-weekdays, 15-minute period and 15 sessions (1.02 minutes for each 25 cm² painful area, analgesic phase, with an anergy 8.0 W, a dose 5 J / cm², a frequency of 25 Hz and total 125 joules) will be applied.
  Interventions: Device: high intensity laser therapy
- exercise+dry needling (Active Comparator): In addition to the exercise program, dry needling (on 3 trigger points on the bilateral trapezius muscle) will be applied to the other 36 randomly selected patients with an acupuncture needle with a size of 0.25x0.25 by the PMR specialist for a total of 6 sessions twice a week for 3 weeks.
  Interventions: Other: dry needle

INTERVENTIONS:
Other: dry needle — dry needling (on 3 trigger points on the bilateral trapezius muscle) will applied to the other 36 randomly selected patients with an acupuncture needle with a size of 0.25x0.25 by the PMR specialist for a total of 6 sessions twice a week for 3 weeks.
  Arms: exercise+dry needling
Device: high intensity laser therapy — High intensity laser therapy (HILT), one of the physical therapy methods, was approved by the FDA in 2002. Its beneficial and versatile effect has been proven in the treatment of many musculoskeletal diseases. In addition to the exercise program, randomly selected 36 case patients + HILT (BTL brand 6000 series, United Kingdom), to the cervical area, for the a period of 3 week-weekdays, 15-minute period and 15 sessions (1.02 minutes for each 25 cm² painful area, analgesic phase, with an anergy 8.0 W, a dose 5 J / cm², a frequency of 25 Hz and total 125 joules) will be applied.
  Arms: exercise+HILT

SUMMARY:
108 myofascial pain syndrome (MPS) diagnosed patients will be randomly divided into 3 groups. To groups; exercise, exercise+high-intensity laser therapy (HILT) and exercise+dry needling will be applied. Visual anolog scale (VAS) scores and neck range of motion (ROM) of the patients before-after treatment will be recorded and will be evaluated statistically.

DETAILED DESCRIPTION:
Myofascial pain syndrome (MPS) is a very common disease in the population that seriously affects the quality of life. Although many modalities are used in its treatment, there is still no common protocol. In this study, the investigators aim to compare the effectiveness of high-intensity laser therapy (HILT), which has been popular in recent years, with exercise and dry needling options that have been used for years.

In our study 108 myofascial pain syndrome (MPS) diagnosed patients will be randomly divided into 3 groups. To groups; exercise, exercise+high-intensity laser therapy (HILT) and exercise+dry needling will be applied. Visual anolog scale (VAS) scores and neck range of motion (ROM) of the patients before-after treatment will be recorded and will be evaluated statistically.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with neck and / or back pain
* diagnosed with MPS
* had a taut band on the trapezius muscle and at least one active trigger point

Exclusion Criteria:

* Diagnosed with fibromyalgia,
* had systemic disease,
* significant cervical disc lesion / radiculopathy / myelopathy,
* had trigger point injection in the last 6 months,
* had neck or shoulder surgery in the year before being included in the study,
* was pregnant,
* received anticoagulant therapy,
* used aspirin in the last three days, and
* with the cognitive dysfunction patients

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Visual anolog scale (VAS) | 10 seconds
  A Visual Analogue Scale (VAS) is a horizontal line, 100 mm in length measurement instrument that tries to measure the amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain.

SECONDARY OUTCOMES:
neck range of motion (ROM) | 3 minutes
  Range of motion (ROM) of the cervical vertebra (flexion, extansion, right-left lateral flexion, right-left rotation) will be measured with goniometre 3 times by a physiotherapist, who does not know the content of the study and mean values will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: emine dundar ahi, assoc prof, Principal Investigator — private medar hospital
Locations (1):
- Private Medar Hospital, Kocaeli, Turkey (Türkiye)

REFERENCES:
- [Derived] Ahi ED, Sirzai H. Comparison of the effectiveness of dry needling and high-intensity laser therapy in the treatment of myofascial pain syndrome: a randomized single-blind controlled study. Lasers Med Sci. 2022 Dec 20;38(1):3. doi: 10.1007/s10103-022-03687-w. PMID 36538189